CLINICAL TRIAL: NCT06120283
Title: A Phase 1a/1b Study Investigating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of the CDK4 Inhibitor BGB-43395, Alone or as Part of Combination Therapies in Patients With Metastatic HR+/HER2- Breast Cancer and Other Advanced Solid Tumors
Brief Title: BGB-43395 Alone or as Part of Combination Therapies in Participants With Breast Cancer and Other Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-43395-101; 2023-506888-34-00 (Registry Identifier: EU CTIS); CTR20243370 (Registry Identifier: ChinaDrugTrials.org)
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor; Advanced Breast Cancer; Metastatic Breast Cancer; Hormone-receptor-positive Breast Cancer; Hormone Receptor Positive Breast Carcinoma; Hormone Receptor Positive Malignant Neoplasm of Breast; HER2-negative Breast Cancer; Hormone Receptor Positive HER-2 Negative Breast Cancer; Non-small Cell Lung Cancer
Keywords: breast cancer; advanced solid tumor; advanced breast cancer; hormone receptor positive breast cancer; HER2-negative breast cancer; Hormone Receptor Positive HER-2 Negative Breast Cancer; BGB-43395; non-small cell lung cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Fulvestrant; Letrozole; elacestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation and Safety Expansion (Experimental): Phase 1a: Sequential cohorts of increasing dose levels of BGB-43395 will be evaluated as monotherapy and in combination with either fulvestrant, letrozole, or elacestrant to assess for safety and tolerability.
  Interventions: Drug: BGB-43395; Drug: Fulvestrant; Drug: Letrozole; Drug: Elacestrant
- Dose Expansion (Experimental): Phase 1b: The recommended dose for expansion (RFDE) for BGB-43395 (in combination with fulvestrant or letrozole) from Phase 1a will be evaluated in HR+ breast cancer and selected tumor-specific cohorts.
  Interventions: Drug: BGB-43395; Drug: Fulvestrant; Drug: Letrozole

INTERVENTIONS:
Drug: BGB-43395 — Planned doses administered orally.
Drug: Fulvestrant — Standard dose administered via intramuscular injection.
Drug: Letrozole — Standard dose administered orally as a tablet.
Drug: Elacestrant — Standard dose administered orally as a tablet.
  Arms: Dose Escalation and Safety Expansion

SUMMARY:
This is a dose escalation and dose expansion study to compare how well BGB-43395, a selective cyclin-dependent kinase 4 (CDK4) inhibitor, works as monotherapy or in combination with fulvestrant, letrozole, or elacestrant in participants with hormone receptor positive (HR+) and human epidermal growth factor 2 negative (HER2-) breast cancer (BC) and other advanced solid tumors. The main purpose of this study is to explore the recommended dosing for BGB-43395.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1a (Dose Escalation) and 1b (Dose Expansion): Participants with histologically or cytologically confirmed advanced, metastatic, or unresectable solid tumors associated with dependency on CDK4, including HR+ breast cancer, ovarian cancer, endometrial cancer, non-small cell lung cancer, and others.
* Phase 1a: Received prior therapy for their condition (if available) and should be refractory to, or intolerant of standard-of-care therapies. In regions where approved and available, participants with HR+ breast cancer must have received at least 2 prior lines of treatment including endocrine therapy and a CDK4/6 inhibitor. For combination with elacestrant, participants must have received at least 1 prior line of treatment for advanced/metastatic disease including prior endocrine therapy and CDK4/6 inhibitor in either the adjuvant or advanced/metastatic setting.
* Phase 1b: Selected tumor cohorts will include HR+/HER2- breast cancer and additional tumor types.
* Phase 1b: Participants with HR+/HER2- breast cancer enrolled in regions where CDK4/6 inhibitors are approved and available must have received at least one line of therapy for advanced disease including endocrine therapy and a CDK4/6 inhibitor. Participants can have received up to 2 lines of prior cytotoxic chemotherapy for advanced disease.
* Stable Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1.
* Female participants with metastatic HR+/HER2- breast cancer must be postmenopausal or receiving ovarian function suppression treatment.
* Adequate organ function without symptomatic visceral disease.

Exclusion Criteria:

* Prior therapy selectively targeting CDK4 (prior CDK4/6 inhibitor therapy is permitted and required in local regions where it is approved and available).
* Known leptomeningeal disease or uncontrolled, untreated brain metastases.
* Any malignancy ≤ 3 years before the first dose of study treatment(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent (eg, resected basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast).
* Uncontrolled diabetes.
* Infection requiring systemic antibacterial, antifungal, or antiviral therapy ≤ 28 days before the first dose of study drug(s), or symptomatic COVID-19 infection.
* Participants with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers with HBV DNA ≥ 500 IU/mL (or ≥ 2500 copies/mL) at screening.
* Participants with active hepatitis C infection.
* Prior allogeneic stem cell transplantation, or organ transplantation.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 60 months
  Number of participants with AEs and SAEs, including findings from physical examinations, electrocardiograms (ECGs), laboratory assessments, and that meet protocol-defined dose-limiting toxicity (DLT) criteria.
Phase 1a: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) of BGB-43395 | Up to approximately 60 months
  MTD is defined as the highest dose evaluated for which estimated toxicity rate is the closest to the target toxicity rate of 28%. MAD is defined as the highest dose administered if MTD is not reached.
Phase 1a: Recommended Dose for Expansion (RDFE) of BGB-43395 | Up to approximately 60 months
  RDFE of BGB-43395 alone or in combination with fulvestrant, letrozole, or elacestrant will be determined based upon the MTD or MAD.
Phase 1b: Objective Response Rate (ORR) | Up to approximately 60 months
  ORR is defined as the percentage of participants who have confirmed complete response (CR) or partial response (PR) assessed by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Phase 1a: ORR | Up to approximately 60 months
  ORR is defined as the percentage of participants who have confirmed CR or PR assessed by the investigator using RECIST v1.1.
Phase 1a and 1b: Duration of Response (DOR) | Up to approximately 60 months
  DOR is defined as the time from the first determination of an overall response per RECIST v1.1 until the first documentation of disease progression or death, whichever occurs first as assessed by the investigator.
Phase 1a and 1b: Time to Response (TTR) | Up to approximately 60 months
  TTR is defined as the time from the date of the first dose of study drugs to the date of the first determination of objective response by the investigator using RECIST v1.1.
Phase 1b: Disease Control Rate (DCR) | Up to approximately 60 months
  DCR is defined as the percentage of participants with best overall response of CR, PR, or stable disease assessed by the investigator using RECIST v1.1.
Phase 1b: Clinical Benefit Rate (CBR) | Up to approximately 60 months
  CBR is defined as the percentage of participants with best overall response of confirmed CR, PR, or stable disease lasting ≥ 24 weeks.
Phase 1b: Progression-Free Survival (PFS) | Up to approximately 60 months
  PFS is defined as the time from the date of the first dose of study drug(s) to the date of the first documentation of progressive disease assessed by the investigator using RECIST v1.1 or death, whichever occurs first.
Phase 1b: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 60 months
  Number of participants with AEs and SAEs, including findings from physical examinations, electrocardiograms (ECGs), and laboratory assessments.
Phase 1a: Observed Plasma Maximum Concentration (Cmax) of BGB-43395 and its metabolite | From Cycle 1 Day 1 up to Cycle 7 Day 1 (each cycle is 28 days)
Phase 1a: Observed Plasma Trough Concentration (Ctrough) of BGB-43395 and its metabolite | From Cycle 1 Day 1 up to Cycle 7 Day 1 (each cycle is 28 days)
Phase 1a: Area under the concentration-time curve (AUC) of BGB-43395 and its metabolite | From Cycle 1 Day 1 up to Cycle 7 Day 1 (each cycle is 28 days)
Phase 1a: Half-life (t1/2) of BGB-43395 and its metabolite | From Cycle 1 Day 1 up to Cycle 7 Day 1 (each cycle is 28 days)
Phase 1b: Plasma concentrations of BGB-43395 and its metabolite | From Cycle 1 Day 1 up to Cycle 5 Day 1 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (63):
- United States (10):
  - Sarah Cannon Research Institute (Scri) At Health One, Denver, Colorado
  - Florida Cancer Specialists and Research Institute, Lake Mary, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Duke Cancer Center, Durham, North Carolina
  - James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Scri Oncology Partners, Nashville, Tennessee
  - Next Oncology, Austin, Texas
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
  - Next Dallas, Irving, Texas
- Australia (8):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Southern Highlands Private Hospital, Bowral, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Macquarie University, North Ryde, New South Wales
  - Townsville University Hospital, Douglas, Queensland
  - Genesiscare St Andrews, Adelaide, South Australia
  - Austin Health, Heidelberg, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
- Brazil (11):
  - Fundacao Pio Xii Hospital de Amor de Barretos, Barretos
  - Hospital Sirio Libanes Brasilia, Brasília
  - Centro de Pesquisas Oncologicas Cepon, Florianópolis
  - Liga Norte Riograndene Contra O Cancer, Natal
  - Fundacao Universidade de Caxias Do Sul Instituto de Pesquisas Em Saude, Petrópolis
  - Hospital Sao Lucas Da Pucrs Uniao Brasileira de Educacao E Assistencia, Porto Algre
  - Instituto Nacional de Cancer, Rio de Janeiro
  - Instituto Dor de Pesquisa E Ensino Hospital Sao Rafael, Salvador
  - Icesp Instituto Do Cancer Do Estado de Sao Paulo Octavio Frias de Oliveira, São Paulo
  - Clinica de Pesquisa E Centro de Estudos Em Oncologia Ginecologica E Mamaria, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
- China (7):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat Sen Memorial Hospital, Sun Yat Sen University (South), Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Centerpudong, Shanghai, Shanghai Municipality
- France (8):
  - Centre de Lutte Contre Le Cancer Institut Bergonie, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Institut Paoli Calmettes, Marseille
  - Institut Curie, Paris
  - Centre Eugene Marquis, Rennes
  - Institut de Cancerologie de Louest, Saint-Herblain
  - Institut Gustave Roussy, Villejuif
- Japan (3):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Shizuoka Cancer Center, Suntogun, Shizuoka
- Malaysia (4):
  - Pulau Pinang Hospital, George Town
  - University Malaya Medical Centre, Kuala Lumpur
  - Sarawak General Hospital, Kuching
  - National Cancer Institute (Institut Kanser Negara), Putrajaya
- The Institute of Oncology, Arensia Exploratory Medicine, Chisinau, Moldova
- New Zealand (2):
  - Harbour Cancer and Wellness, Auckland
  - Nzcr Christchurch, Christchurch
- South Korea (8):
  - Seoul National University Bundang Hospital, BundangGu SeongnamSi, Gyeonggi-do
  - Gachon University Gil Medical Center, NamdongGu, Incheon Gwang'yeogsi
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St Marys Hospital, SeochoGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Korea University Anam Hospital, SeongbukGu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, SongpaGu, Seoul Teugbyeolsi
- Srinagarind Hospital (Khon Kaen University), Muang, Thailand

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/